CLINICAL TRIAL: NCT02909816
Title: Adverse Event Risk Assessment in the Use of Nitrous Oxide for Pediatric Dental Patients
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Frederic COURSON, PhD, DDS, Assistance Publique - Hôpitaux de Paris
Other Study IDs: MEOPA
Record Dates: First submitted 2016-09-09; First posted 2016-09-21 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Dental Carie; Orthodontics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective was to assess adverse event risk in the use of Nitrous Oxide for Pediatric Dental Patients. The investigators performed a multicenter observational study. The investigators included patients aged 1 to 18 years and who have already failed dental care because of non-cooperation; they could be with mental or cognitive disabilities and could have sedative premedication. The investigators performed any type of dental care With the Use of Nitrous Oxide/Oxygen Sedation. The primary outcome was vomiting assessed during or after dental care.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 18 years
* Use of nitrous oxide/oxygen analgesia/anxiolysis
* Any type of dental care

Exclusion Criteria:

* Use of midazolam
* Use of general anesthesia

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Patients under 18 years
  * Patients who have already failed dental care because of non-cooperation
  * Patients with or without mental or cognitive disabilities (regardless of type)
  * Patients with or without sedative premedication
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
occurrence of vomiting | from the beginning of Nitrous Oxide/Oxygen administration up to half an hour after the end of dental treatment

CONTACTS AND LOCATIONS:
Overall Officials: Violaine Smaïl-Faugeron, PhD, DDS, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Violaine Smaïl-Faugeron, Paris, France

IPD SHARING:
Plan to Share IPD: No